CLINICAL TRIAL: NCT06433869
Title: Multi-arm, Phase II Clinical Study of Intraperitoneal Injection of Recombinant Human Tumor Necrosis Factor, Bevacizumab Monoclonal Antibody, and Serplulimab for the Treatment of Malignant Ascites Patients With Standard Therapy Failure
Brief Title: The Efficacy of Bevacizumab and Serplulimab Combined With Recombinant Mutant HumanTumor Necrosis Factor(rmhTNF-NC) in the Treatment of Malignant Ascites
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, Director, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPPMS-001
Record Dates: First submitted 2024-04-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Malignant Ascites
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Bevacizumab; recombinant human tumor necrosis factor-binding protein-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Treat the malignant ascites by local intraperitoneal injection of PD-1 inhibitor and bevacizumab
  Interventions: Drug: serplulimab; Drug: Bevacizumab
- Group B (Experimental): Treat the malignant ascites by local intraperitoneal injection of PD-1 inhibitor and rmhTNF-NC
  Interventions: Drug: serplulimab; Drug: rmhTNF-NC
- Group C (Experimental): Treat the malignant ascites by local intraperitoneal injection of PD-1 inhibitor, rmhTNF-NC and bevacizumab
  Interventions: Drug: serplulimab; Drug: Bevacizumab; Drug: rmhTNF-NC

INTERVENTIONS:
Drug: serplulimab — Additional intraperitoneal injection of bevacizumab or rmhTNF-NC is added to the PD-1 inhibitor.
  Other Names: PD-1 inhibitor
Drug: Bevacizumab — Intraperitoneal injection of bevacizumab is added to PD-1 inhibitor or rmhTNF-NC.
  Arms: Group A; Group C
Drug: rmhTNF-NC — Intraperitoneal injection of rmhTNF-NC is added to PD-1 inhibitor or bevacizumab.
  Other Names: recombinant human tumor necrosis factor
  Arms: Group B; Group C

SUMMARY:
1. More than half of peritoneal metastases are from digestive tract. Peritoneal metastasis has poor prognosis, poor treatment response and limited means.
2. rmhTNF-NC or bevacizumab are effective in the treatment of malignant pleuroabdominal effusion.

3, There is increasing evidence that PD-1/PD-L1 inhibitors in combination with vascular endothelial growth factor receptor (VEGFR) inhibitors have a complementary mechanism of action: VEGF pathway inhibitors normalize blood vessels in tumors and promote immune cell maturation and infiltration, thus playing a synergistic role with ICIs. The strategy of systemic immunotherapy combined with antivascular therapy has been confirmed by several large phase III clinical trials such as IMbrave-150. Basic studies have confirmed that uncontrolled tumor vessels in peritoneal metastasis and malignant ascites microenvironment also play an important role in promoting disease progression. Therefore, this project intends to explore the treatment of malignant abdominal effusion by local intraperitoneal injection of bevacizumab and PD-1 on the basis of rmhTNF-NC

DETAILED DESCRIPTION:
GROUP A: serplulimab(PD-1 inhibitor)+bevacizumab GROUP B: serplulimab+rmhTNF-NC GROUP C: serplulimab+bevacizumab+rmhTNF-NC

serplulimab(100mg,ip,D1、D15) bevacizumab(100mg,ip,D1、D15) rmhTNF-NC(300IU/time,ip,D1、D4、D7、D10)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, gender unlimited;
* Malignant ascites confirmed by histology or cytology as originating from digestive system tumors (malignant confirmed by ascites cytology or clinically diagnosed as peritoneal metastases by imaging and symptoms);
* Patients with more than a moderate amount of abdominal fluid, who have failed initial treatment or have been treated with conventional chemotherapy drugs and/or biological response modulators intravenously. Moderate ascites is defined as:

  * B ultrasound examination of ascites ≥3cm in lying position;
  * Accompanied by clinical symptoms (chest tightness, shortness of breath, abdominal distension and discomfort, which were judged by researchers to be related to abdominal fluid accumulation);
* ECOG physical status is 0-2;
* Expected survival time >3 months;
* Cardiopulmonary function is basically normal;
* For adequate organ function, subjects must meet the following laboratory criteria:

  * Peripheral blood imaging: WBC≥4.0×109/L, PLT≥80×109/L, Hb≥90g/L;
  * Renal function: serum creatinine ≤2×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥40 ml/min;
  * Liver function: total bilirubin ≤1.5× upper limit of normal value (ULN); Or total bilirubin >ULN but direct bilirubin ≤ ULN; Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
  * Good coagulation function, defined as International standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
* Thyroid stimulating hormone (TSH) ≤ULN; If abnormal, T3 and T4 levels and clinical manifestations should be investigated, and comprehensive assessment of non-acute activity can be included;
* Non-surgical sterilization or female patients of reproductive age who are required to use a medically approved contraceptive method (such as an IUD, contraceptive pill or condom) during the study treatment period and for 6 months after the end of the study treatment period; Women of reproductive age who were not surgically sterilized had to be negative for serum or urine HCG within 7 days prior to study enrollment. And must be non-lactation period; For men whose partners are women of childbearing age, effective contraception should be used during the trial and within 6 months after the last administration of the study drug;
* Voluntarily enrolled in this study, with good compliance, signed written informed consent, and able to cooperate with follow-up observation.

Exclusion Criteria:

* History of allergy to tumor necrosis factor and its derivatives, bevacizumab analogues, and Serplulimab;
* Malignant diseases other than digestive tract neoplasms were diagnosed within 5 years prior to initial administration (excluding radical basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or carcinoma in situ after radical resection);
* Received any other investigational drug therapy or participated in an interventional clinical investigator within 7 days prior to initial dosing; Or received anti-tumor drug treatment (including Chinese herbal medicine with anti-tumor indication) within 7 days prior to the first use of the study drug;
* Pregnant or lactating women, women of childbearing age who did not want to use contraception during the study period; Or the man is unwilling to use effective contraception during treatment and during the following 1 year;
* Significant damage to the function of important organs;
* Patients with obvious bleeding tendency;
* Clinically significant or uncontrolled heart disease, including unstable angina pectoris, acute myocardial infarction within 6 months prior to first dosing, New York Heart Association Class III/IV congestive heart failure, and uncontrolled arrhythmia (in subjects who are allowed to wear a pacemaker or have atrial fibrillation and have a well-controlled heart rate);
* Presence of ECG changes or medical history that investigators consider clinically significant; Screening QTcF interval >480 ms, subjects with indoor block (QRS interval >120 ms) can use JTc interval instead of QTc interval (if JTc is used instead of QTc, JTc must be ≤340 ms);
* Uncontrolled hypertension, systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy;
* Severe acute infection that is not under control; The patient is having fever (> 38℃), or has suppurative and chronic infection, and the wound is prolonged and does not heal;
* Patients with encapsulated abdominal effusion confirmed by imaging; A definite diagnosis of abdominal infection;
* Persons infected with acute or chronic active hepatitis B or hepatitis C, hepatitis B virus (HBV) DNA>2000IU/ml or 104 copies /ml; Hepatitis C virus (HCV) RNA> 103 copies /ml; Hepatitis B surface antigen (HbsAg) and anti-HCV antibodies were both positive. After nucleotide antiviral therapy, those who were lower than the above criteria could be included in the group. A known history of human immunodeficiency virus (HIV) infection or a confirmed positive immunotest result;
* Patients with obvious evidence of bleeding tendency or history within 3 months prior to enrollment (hemorrhage >30 mL within 3 months, hematemesis, stool, and blood in the stool), hemoptysis (>5 mL fresh blood within 4 weeks); People with a history of inherited or acquired bleeding or coagulation disorders. Have clinically significant bleeding symptoms or definite bleeding tendency within 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.; Arterial or venous thrombotic disease was present 6 weeks before enrollment;
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
* Had a major surgical procedure (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study therapy or expected to require major surgery during study therapy;
* Complications of toxicity and/or major surgery have not fully recovered before starting treatment;
* Women who are pregnant or nursing, or who are expected to become pregnant or give birth during the study period from screening visits to completion of safety follow-up visits (male subjects to 90 days after the last dosing);
* Radiotherapy was received within 4 weeks prior to the first administration of the study drug. Subjects must have fully recovered from radiation-related toxicities without the need for corticosteroid therapy, confirming the rule out of radiation pneumonia. For palliative radiotherapy for non-CNS disease, a 2-week washout period is allowed;
* Patients with uncontrollable neurological, mental illness or mental disorder, poor compliance, unable to cooperate with and describe the response to treatment; Patients with uncontrolled primary brain tumor or central nervous metastases, with obvious cranial hypertension or neuropsychiatric symptoms;
* There are other conditions that researchers consider inappropriate to participate in this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate of ascites | 2 months
  Defined as the percentage of patients achieving CR or PR according to the WHO criteria detected by ultrasound.

SECONDARY OUTCOMES:
Duration of ascites relief | 1 years
  Time since first CR or PR to PD
Ascites control rate | 2 months
  percentage of patients achieving CR, PR and SD.
Incidence of Treatment-Emergent Adverse Events | 2 months
  Adverse events according to the NCI CTCAE 5.0
The score of chronic abdominal effusion function scale changed | 2 months
  Measured by FACIT-AI,score range 1 to 5, higher scores mean a better

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer center of SunYat-sen University, Guangzhou, Guangdong
  - Zhang Dongsheng, Guangzhou

IPD SHARING:
Plan to Share IPD: Undecided